CLINICAL TRIAL: NCT04482413
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of AstroStem, Autologous Adipose Tissue Derived Mesenchymal Stem Cells, in Patients With Alzheimer's Disease
Brief Title: Study to Evaluate the Safety and Efficacy of AstroStem in Treatment of Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nature Cell Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AST-ADP2-US02
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Treatment group will be administered via intravenously AstroStem which consists of two syringes and each syringe contains 2.0 x 10^8 cells / 20 mL of saline with 30% auto-serum.
  Interventions: Drug: AstroStem
- Placebo Control (Placebo Comparator): Placebo control group will receive AstroStem Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AstroStem — Treatment group receive AstroStem(Autologous adipose tissue derived mesenchymal stem cells, AdMSCs) every 4 weeks from Week 0 to Week 36.
  Arms: Treatment
Drug: Placebo — Placebo control group receive 20 mL of Saline and auto serum every 4 weeks from Week 0 to Week 36.
  Other Names: AstroStem Placebo
  Arms: Placebo Control

SUMMARY:
This is a phase 2b randomized, double-blind, Placebo-controlled study with 2 treatment arms, to compare the efficacy and safety of AstroStem vs. Placebo treatment in patients with mild Alzheimer's Disease(AD). Eligible patients diagnosed with AD within one year of the start of treatment will be enrolled. Patients who are randomized into the treatment group will be administered via intravenously AstroStem every 4 weeks from Week 0 to Week 36. On the other hand, patients who are randomized into the placebo control group will receive Placebo every 4 weeks from Week 0 to Week 36. After the final administration, patients will be scheduled for two follow-up visits, at Weeks 44 and 52, to assess efficacy and safety endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 50 and above at the time of signing the Informed Consent Form
* Patients who can understand and provide written informed consent (assent)
* Patients who have a diagnosis of probable mild Alzheimer's Disease(AD) according to the National Institute of Neurological and Communicative Disorders and Stroke; Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria within one year of the start of treatment
* Patients who have an MMSE Score of 20 to 24 at screening
* Patients who have a Clinical Dementia Rating (CDR)-Global Score of 0.5 to 1 at baseline
* Patients who have any FDA-approved AD medication (donepezil, galantamine, memantine, rivastigmine or any combination) since their AD diagnosis receiving a stable dose of medical teratment for at least 12 weeks prior to Screening and were to stay on a stable dose during the study
* Patients who have one (or more) identified adult caregiver (study partner) who is able to read, understand, and speak the designated language at the study site; who either lives with the subject or sees the subject for ≥2 hours/day ≥4 days/week; and who agrees to accompany the subject to each study visit and to participate in the subject's clinical assessments
* Patients who have a diagnosis of probable mild AD according to Amyloid PET scan at screening

Exclusion Criteria:

* Female patients who are pregnant, nursing, or of childbearing potential while not practicing effective contraception
* Patients who have signs of delirium
* Patients who have had a cortical stroke within the preceding 2 years
* Patients who have a prolonged QTc interval at screening; >450 msec for males or >470 msec for females
* Patients who have a diagnosis of severe white matter hyperintensity (WMH), which is defined as ≥25mm of the deep white matter and ≥10mm of the periventricular capping/banding in lengths
* Patients who have a diagnosis of dementia or cause of cognitive impairment other than AD
* Patients who have a significant abnormal result in laboratory tests, in the opinion of the investigator
* Patients who have participated in any investigational drug, stem cell therapy, or device trial within the previous 3 months at screening
* Patients with any current psychiatric diagnosis other than AD if, in the judgment of the investigator, the psychiatric disorder or symptom is likely to confound interpretation of drug effect, affect cognitive assessments, or affect the subject´s ability to complete the study
* Patients who are known to have autosomal dominant mutation-associated presenile AD
* Patients who show signs of Acquired Immunodeficiency Syndrome (AIDS), Hepatitis B Virus (HBV), Hepatitis C (HCV), Venereal Disease Research Laboratory (VDRL)
* Patients who have any conditions that would contraindicate an MRI, such as the presence metallic objects in the eyes, skin, or heart
* Patients who have >4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis, or evidence of a prior microhemorrhage as assessed by MRI
* Patients who have history of malignant cancer within the last 5 years (The following is a partial list of conditions that are permissible for study entry: non-metastatic basal and/or squamous cell carcinoma of the skin, in situ cervical, or non-progressive prostate cancer)
* Patients who have suspected active lung disease based on chest X-ray
* Patients who are hypersensitive to fetal bovine serum or penicillin
* Patients who are currently using immunosuppressants, cytotoxic drug, corticosteroids or similar steroidal anti-inflammatory medication (e.g., Prednisone) on a regular basis (exceptions allowed include; regular use of steroidal nasal sprays, topical steroids, and estrogen-replacement therapy)
* Patients for whom the investigator judges the liposuction may cause a problem

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
SUVR (Standard Uptake Value Ratio) | Baseline and 52 Weeks
  Standard Uptake Value Ratio (SUVR) of the Amyloid PET scan

SECONDARY OUTCOMES:
CDR-SB score (Clinical Dementia Rating Sum of Boxes) | Baseline and 52 Weeks
  Changes of CDR-SOB from baseline at Week 52 Score range: 0-18.0 0 = normal, 0.5-4.0 = questionable cognitive dementia, 4.5-9.0 = mild dementia, 9.5-15.5 = moderate dementia, and 16.0-18.0 = severe dementia
ADAS-Cog-11 score (Alzheimer's Disease assessment Scale-Cognitive Subscale (11 items)) | Baseline and 52 Weeks
  Change of ADAS-Cog (Alzheimer's Disease Assessment Scale-cognitive subscale) from Baseline at Week 52 Score range: 0-70 A score of 70 represents the most severe impairment and 0 represents the least impairment
MMSE (Mini-mental status examination) | Baseline and 52 Weeks
  Change from baseline to Week 52 in the Mini-mental status examination (MMSE) score. The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
ADCS-ADL-MCI (Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory) | Baseline and 52 Weeks
  Change from baseline to Week 52 in the ADCS-ADl MCI 0-53 A score of 0 represents the most severe impairment and 53 represents the least impairment
C-SSRS (Columbia Suicide Severity Rating Scale) | Baseline and 52 Weeks
  Change from baseline to Week 52 in the Columbia Suicide Severity Rating Scale (C-SSRS) score. The suicidal ideation severity subscale ranges from 1 to 5 (with higher number indicating more severe ideation). The intensity of ideation subscale includes 5 questions each one ranging from 1 to 5 (with higher number indicating more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
NPI (Neuropsychiatric Inventory) | Baseline and 52 Weeks
  Change from baseline to Week 52 in the Neuropsychiatric Inventory (NPI) score. The NPI is a structured interview with a caregiver or qualified study partner (defined as having direct contact > 2 days/week) that evaluates both presence and severity of 12 neuropsychiatric features which include: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability, lability, apathy, aberrant motor behavior, night-time behavior, and appetite/ eating changes. If the response to the domain question is "No", the informant goes to the next question. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale ranging from 1 to 3 (mild to severe).
Treatment related Adverse Events | Baseline and 52 Weeks
  Number of subjects with treatment related adverse events as assessed by analysis of adverse events including symptoms, and abnormal findings on physical examination, vital signs, ECG, and standard laboratory examination results

IPD SHARING:
Plan to Share IPD: Undecided